CLINICAL TRIAL: NCT01696825
Title: COMPARISON OF ABSORPTION OF VAGINAL DIAZEPAM USING DIFFERENT DELIVERY SYSTEMS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Jason Gilleran (Other)
Responsible Party: Sponsor-Investigator, Jason Gilleran, Physician, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-182
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Metabolism, Drug
MeSH Terms: interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diazepam Tablet, 5 mg, Vaginal (Experimental)
  Interventions: Drug: Diazepam tablet, 5 mg, vaginal
- Diazepam Suppository, 5 mg, Vaginal (Experimental)
  Interventions: Drug: Diazepam Suppository, 5 mg, vaginal
- Diazepam Cream, 5 mg, Vaginal (Experimental)
  Interventions: Drug: Diazepam Cream, 5 mg, Vaginal
- Diazepam Tablet, 5 Mg, Oral (Active Comparator)
  Interventions: Drug: Diazepam tablet, 5 mg, vaginal; Drug: Diazepam Suppository, 5 mg, vaginal; Drug: Diazepam Cream, 5 mg, Vaginal

INTERVENTIONS:
Drug: Diazepam tablet, 5 mg, vaginal — Diazepam tablet, 5 mg, moistened and inserted vaginally
  Other Names: Valium
  Arms: Diazepam Tablet, 5 Mg, Oral; Diazepam Tablet, 5 mg, Vaginal
Drug: Diazepam Suppository, 5 mg, vaginal — Compounded diazepam 5 mg suppository administered vaginally
  Other Names: Valium
  Arms: Diazepam Suppository, 5 mg, Vaginal; Diazepam Tablet, 5 Mg, Oral
Drug: Diazepam Cream, 5 mg, Vaginal — Compounded diazepam cream, 5 mg, inserted vaginally
  Other Names: Valium
  Arms: Diazepam Cream, 5 mg, Vaginal; Diazepam Tablet, 5 Mg, Oral

SUMMARY:
The purpose of this study is to determine which of three delivery systems of vaginal diazepam have the best systemic absorption, measured by serum diazepam levels. The three delivery systems are: moistened tablet, suppository or cream. Additionally the study will compare the side effects and absorption of vaginal diazepam with oral diazepam. Vaginal diazepam is used off-label vaginally to relax pelvic floor muscles and reduce pelvic pain caused from pelvic floor dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Premenopausal women > age 18
* Able to provide urine and serum samples during the time period

Exclusion Criteria:

* Current use of benzodiazepines in any form. If history of benzodiazepine use, must not have taken for one week prior to study screening and enrollment
* Pregnancy
* Concomitant use of any narcotic drug, ethanol, or any illicit drug use during the study period that could be deemed unsafe in combination with benzodiazepine medication use as judged by the investigators.
* Any evidence of vaginitis on wet mount slide
* Postmenopausal
* Subject with any other vaginal epithelial disorder that could affect absorption of medication as deemed by the investigators.
* Any indication/condition/medication that the investigators identify as contraindicated in conjunction with diazepam.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Serum diazepam levels measured over time | Baseline then 2 hours, 4 hours and 8 hours post-medication administration

SECONDARY OUTCOMES:
Side effects observed with each of three types of vaginal diazepam | Baseline and 2 hours, 4 hours and 8 hours post medication administration

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gilleran, MD, Principal Investigator — Corewell Health East
Locations (1):
- Women's Urology Center, William Beaumont Hospital, Royal Oak, Michigan, United States